CLINICAL TRIAL: NCT01200589
Title: Phase III Randomized, Open Label Study of Single Agent Ofatumumab Vs. Single Agent Rituximab in Indolent B-Cell Non Hodgkin Lymphoma Relapsed After Rituximab-Containing Therapy
Brief Title: Single Agent Ofatumumab Vs. Single Agent Rituximab in Indolent B-Cell Non Hodgkin Lymphoma Relapsed After Rituximab-Containing Therapy
Acronym: HOMER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study stopped due to futility.
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 113676
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-04

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Randomized trial; Ofatumumab; Rituximab; Indolent B-Cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ofatumumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Ofatumumab (Experimental): Four weekly doses of single agent ofatumumab (1000 mg), followed by ofatumumab (1000 mg) every two months for four additional doses.
  Interventions: Biological: Ofatumumab
- Arm B: Rituximab (Active Comparator): Four weekly doses of single agent rituximab (375 mg/m2), followed by rituximab (375 mg/m2) every two months for four additional doses.
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: Ofatumumab — liquid concentrate for solution for infusion in glass vials containing 50 mL of solution at a concentration of 20mg/ml to provide 1000 mg per vial.
  Other Names: Arzerra
  Arms: Arm A: Ofatumumab
Biological: Rituximab — sourced locally from commercial stock
  Other Names: Mabthera; Rituxan
  Arms: Arm B: Rituximab
Biological: Ofatumumab — Four weekly doses of single agent ofatumumab (1000 mg), followed by ofatumumab (1000 mg) every two months for four additional doses.
  Other Names: Arzerra
  Arms: Arm A: Ofatumumab
Biological: Rituximab — Four weekly doses of single agent rituximab (375 mg/m2), followed by rituximab (375 mg/m2) every two months for four additional doses.
  Other Names: Mabthera; Rituxan
  Arms: Arm B: Rituximab

SUMMARY:
This was a multi-center, parallel, active comparator controlled, open-label, randomized (1:1) phase III study of single agent ofatumumab compared to single agent rituximab in subjects with rituximab-sensitive indolent B-cell non hodgkin lymphoma that has relapsed at least 6 months after completing treatment with single agent rituximab or a rituximab-containing regimen. Subjects must have attained a Complete Response or Partial Response to their last prior rituximab containing therapy lasting at least six months beyond the end of rituximab therapy. Subjects were to receive four weekly doses of single agent ofatumumab (1000 mg) or rituximab (375 mg/m2), followed by ofatumumab (1000 mg) or rituximab (375 mg/m2) every 2 months for four additional doses. Therefore, subjects were to receive a total of eight doses of anti-CD20 antibody over 9 months. Subjects were evaluated for response after completion of the first four doses of therapy, after six doses of therapy, and after completion of study therapy. Subjects were to be followed until the end of the designated follow-up period (total study duration of 200 weeks) or until they meet the withdrawal criteria.

The primary objective of the study OMB157D 2303 was to demonstrate the efficacy of Arzerra based on the primary endpoint (Progression-free survival (PFS) as assessed by the IRC) in patients with Indolent B-cell Non-Hodgkin's Lymphoma Relapsed After Rituximab-Containing Regimen.

The Independent Data Monitoring Committee (IDMC) met on November 22, 2015 and recommended the termination of the study due to futility (cut-off date = 12Jun2015). The IDMC reviewed analyses results for progression free survival (PFS), overall response rate (ORR), and overall survival (OS). Novartis accepted this recommendation and the study was closed.

Final analysis was performed (cut-off date =19 Dec 2016). As the study was stopped for futility, the primary objective was not met and some secondary endpoints, supportive of primary objective (Duration of Response (DOR), time to next therapy, and pharmacokinetics) were removed as secondary end points.

ELIGIBILITY:
Inclusion Criteria:

1. Indolent NHL subtypes defined according to World Health Organization guidelines:

   1. Follicular lymphoma Grades 1, 2, 3 A
   2. Small lymphocytic lymphoma (SLL)
   3. Marginal zone lymphoma
   4. Lymphoplasmacytic lymphoma
2. Rituximab-sensitive iNHL, defined as a partial or complete response to their last prior treatment with rituximab or a rituximab-containing regimen lasting at least 6 months following completion of rituximab treatment.
3. Relapse or disease progression following response to prior rituximab-based therapy, as defined by 2007 RRCML criteria, which requires therapy.
4. Radiographically measurable disease, defined as: 2 or more clearly demarcated lesions/nodes with a long axis >1.5 cm and short axis ≥1.0cm. OR 1 clearly demarcated lesion/node with a long axis >2.0 cm and short axis ≥1.0cm.
5. ECOG Performance Status of 0, 1, or 2.
6. Age ≥18 years.
7. Life expectancy of at least 6 months in the opinion of the investigator.
8. The patient or their legally acceptable representative must be capable of giving written informed consent prior to performing any study-specific tests or procedures.
9. All prior treatment related non-hematologic toxicities (with the exception of alopecia) must have resolved to CTCAE (Version 4.0) ≤ Grade 2 at the time of randomization.
10. One or more of the following indications for treatment:

    1. Cytopenias
    2. One or more of the following lymphoma-related symptoms:

       * Night sweats without signs of infection
       * Unintentional weight loss (10% within the previous 6 months)
       * Recurrent, unexplained fever of greater than 100.5F (38C) without signs of infection
       * Fatigue which interferes with the patient's quality of life
    3. Progressive or massive lymphadenopathy OR
    4. Progressive or massive organomegaly French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

1. Previous treatment with ofatumumab.
2. Previous anti-CD20 radioimmunotherapy (RIT) or non-rituximab anti-CD20 therapy (such as obinutuzumab) within 6 months prior to randomization. Patients who have received previous anti-CD20 RIT or non-rituximab anti-CD20 therapy (such as obinutuzumab) must have attained a partial or complete response lasting at least 6 months, and must have recovered from any hematologic or other toxicity.
3. Previous autologous stem cell transplantation within 6 months prior to randomization.
4. Previous allogeneic stem cell transplantation.
5. Previous anti-lymphoma monoclonal antibody therapy (excluding anti-CD20 therapy and anti-CD20 RIT), chemotherapy, glucocorticoid, or other systemic therapy for lymphoma within 3 months prior to randomization.
6. Current or previous participation in the treatment phase of another interventional clinical study within 4 weeks prior to randomization. Patients may continue in the follow-up phase of another interventional clinical study, but may not have undergone any treatment on the other study within 4 weeks prior to randomization.
7. Current or previous other malignancy within 2 years prior to randomization. Subjects who have been free of malignancy for at least 2 years, or have a history of completely resected non-melanoma skin cancer or successfully treated carcinoma in situ, are eligible.
8. Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis, active Hepatitis C, and known HIV disease. All HIV-positive patients are excluded from this study, regardless of whether they have an Acquired Immunodeficiency Syndrome (AIDS) defining disease and/or are on antiviral therapy. Prophylactic antiviral and/or antibacterial antibiotics to prevent recurrence of previous infections are permitted.
9. Clinically significant cardiac disease as judged by the investigator including unstable angina, acute myocardial infarction within 6 months prior to randomization, uncontrolled congestive heart failure, and uncontrolled arrhythmia. Subjects with congestive heart disease or arrhythmias such as atrial fibrillation whose cardiac disease is well controlled on a stable medical regimen are eligible.
10. Other significant concurrent, uncontrolled medical conditions including, but not limited to, renal, hepatic, autoimmune, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which, in the investigator's opinion, will impact study participation.
11. Screening laboratory values:

    1. Neutrophils < 1.5 x 10^9/L (unless due to iNHL involvement of the bone marrow)
    2. Platelets < 50 x 10^9/L (unless due to iNHL involvement of the bone marrow)
    3. ALT or AST > 3 x ULN
    4. Alkaline phosphatase > 1.5 x ULN (unless due to lymphoma or a non-malignant, non-hepatic cause such as Paget's disease)
    5. Total bilirubin > 1.5 x ULN (unless due to lymphoma or isolated, predominantly indirect hyperbilirubinemia due to Gilbert's syndrome)
12. Known or suspected inability to fully comply with study protocol
13. Because the effects of ofatumumab on fetuses and nursing infants are not known, the following are ineligible for study entry:

    1. Lactating women.
    2. Women with a positive pregnancy test at study entry.
    3. Men with partners of childbearing potential and women of childbearing potential who are not willing to use adequate contraception from study entry through one year following last treatment dose. (Adequate contraception is defined as abstinence, oral hormonal birth control, hormonal birth control injections, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, intrauterine device, and male partner sterilization if male partner is the sole partner for a female subject. The double barrier method can be used in regions where considered acceptable and adequate, defined as condom or occlusive cap plus spermicidal agent).
14. Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones).
15. Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the subject will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2010-10-11 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (132):
- United States (66):
  - Novartis Investigative Site, Anchorage, Alaska
  - Novartis Investigative Site, Gilbert, Arizona
  - Novartis Investigative Site, Hot Springs, Arkansas
  - Novartis Investigative Site, Greenbrae, California
  - Novartis Investigative Site, Monterey, California
  - Novartis Investigative Site, Pleasant Hill, California
  - Novartis Investigative Site, Rancho Mirage, California
  - Novartis Investigative Site, Salinas, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Pablo, California
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, New Milford, Connecticut
  - Novartis Investigative Site, Torrington, Connecticut
  - Novartis Investigative Site, Lakeland, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Pembroke Pines, Florida
  - Novartis Investigative Site, Port Saint Lucie, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Macon, Georgia
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Evanston, Illinois
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Quincy, Illinois
  - Novartis Investigative Site, Skokie, Illinois
  - Novartis Investigative Site, Anderson, Indiana
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Ames, Iowa
  - Novartis Investigative Site, Mount Sterling, Kentucky
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, Shreveport, Louisiana
  - Novartis Investigative Site, Waterville, Maine
  - Novartis Investigative Site, Silver Spring, Maryland
  - Novartis Investigative Site, Grand Rapids, Michigan
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Columbia, Missouri
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Saint Joseph, Missouri
  - Novartis Investigative Site, Springfield, Missouri
  - Novartis Investigative Site, Bozeman, Montana
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Lake Success, New York
  - Novartis Investigative Site, Mount Kisco, New York
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Bismarck, North Dakota
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Danville, Pennsylvania
  - Novartis Investigative Site, Ephrata, Pennsylvania
  - Novartis Investigative Site, Lancaster, Pennsylvania
  - Novartis Investigative Site, Willow Grove, Pennsylvania
  - Novartis Investigative Site, Chattanooga, Tennessee
  - Novartis Investigative Site, Germantown, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Fort Sam Houston, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Ogden, Utah
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Fredericksburg, Virginia
  - Novartis Investigative Site, Kennewick, Washington
  - Novartis Investigative Site, Kirkland, Washington
  - Novartis Investigative Site, Mount Vernon, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Sequim, Washington
  - Novartis Investigative Site, Spokane, Washington
- Belgium (6):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Wilrijk
- Brazil (8):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Betim, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, Jaú, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Rio de Janeiro
- Bulgaria (4):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (4):
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- China (5):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Czechia (4):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Ostrava
  - Novartis Investigative Site, Prague
- France (6):
  - Novartis Investigative Site, Boulogne-sur-Mer
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Pessac
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Szeged
- Japan (7):
  - Novartis Investigative Site, Aichi
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Miyagi
  - Novartis Investigative Site, Nagasaki
  - Novartis Investigative Site, Saitama
  - Novartis Investigative Site, Tochigi
  - Novartis Investigative Site, Tokyo
- Peru (3):
  - Novartis Investigative Site, Miraflores, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, Lima
- Novartis Investigative Site, San Juan, Puerto Rico
- Slovakia (3):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Martin
- South Africa (4):
  - Novartis Investigative Site, Parktown, Gauteng
  - Novartis Investigative Site, Athlone Park, Amanzimtoti
  - Novartis Investigative Site, Port Elizabeth
  - Novartis Investigative Site, Saxonwold, Johannesburg
- South Korea (2):
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Seoul
- Ukraine (5):
  - Novartis Investigative Site, Donetsk
  - Novartis Investigative Site, Kyiv
  - Novartis Investigative Site, Lviv
  - Novartis Investigative Site, Makiivka
  - Novartis Investigative Site, Simferopil

REFERENCES:
- [Derived] Maloney DG, Ogura M, Fukuhara N, Davis J, Lasher J, Izquierdo M, Banerjee H, Tobinai K. A phase 3 randomized study (HOMER) of ofatumumab vs rituximab in iNHL relapsed after rituximab-containing therapy. Blood Adv. 2020 Aug 25;4(16):3886-3893. doi: 10.1182/bloodadvances.2020001942. PMID 32810220

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1 ratio to Ofatumumab or Rituximab.
Groups:
- Ofatumumab: Four weekly doses of single agent ofatumumab 1000 mg by intravenous (i.v.) infusion, followed by ofatumumab 1000 mg i.v. every two months for four additional doses.
- Rituximab: Four weekly doses of single agent rituximab 375 mg/m2 i.v., followed by rituximab 375 mg/m2 i.v. every two months for four additional doses.
Period: Overall Study
Arm/Group | Ofatumumab | Rituximab
Started | 219 | 219
Intent-to-treat (ITT) Analysis Set | 219 | 219
Safety Set | 217 | 218
Completed | 29 | 30
Not Completed | 190 | 189
Not completed — Withdrawal by Subject | 13 | 11
Not completed — Physician Decision | 2 | 2
Not completed — Lost to Follow-up | 5 | 4
Not completed — Study terminated | 170 | 172

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ofatumumab | Rituximab | Total
Number analyzed (Participants) | 219 | 219 | 438
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (11.27) | 60.7 (11.84) | 60.8 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 109 | 224
  Male | 104 | 110 | 214

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) - Number of Participants With PFS Events
Description: Disease response assessed by modified 2007 Revised Response Criteria for Malignant Lymphoma. Nodal disease, PD: 1)prev. normal node (<=1.5cm x <=1.0cm) that incr. to >2.0 x ≥1.5cm; 2)≥50% incr. from nadir product of perpendicular diameter (PPD) of any prev. involved node with long axis >1.5cm at baseline (BL) (must incr. by ≥0.5mm & to >2.0cm) OR ≥50% incr. from nadir in long axis of any prev. inv. node with long axis of >1.5cm at BL (long axis must incr. by ≥0.5mm & to >2.0cm); or 3)≥50% incr. from nadir in the sums of prod. of diameters (SPD) of target nodes & ≥1 node with long axis >1.5cm. Extranodal, PD 1)any new lesion >2.0 x ≥1.5cm not attributed to non-lymphoma causes; 2)≥50% incr. from nadir PPD of any targ. les. & >5mm incr. in either axis & les. must measure >1.5cm x ≥1.5cm OR ≥50% incr. from nadir in long axis of any targ. les. & >5mm incr. in either axis & les. must measure >1.5cm x ≥1.5cm; or 3)≥50% incr. from nadir in SPD of targ. nodes & ≥1 node with long axis >1.5cm.
Time Frame: 200 weeks
Population: The Intent-to-treat (ITT) analysis set, comprised of all randomized participants, was analyzed.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Rituximab
Number analyzed (Participants) | 219 | 219
Participants | 114 | 117
Statistical Analysis 1: Comparison: Ofatumumab vs Rituximab; Test type: Superiority or Other; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.89 to 1.49]

2. Secondary Outcome: Number of Participants With Complete Response (CR)
Description: Complete response was assessed according to modified 2007 Revised Response Criteria for Malignant Lymphoma (RRCML) and defined as follows: 1) complete disappearance of all detectable clinical evidence of disease (all target nodes regressing to <=1.5cm in the long axis and all non-target lesions being normal in size by imaging) and disease-related symptoms if present before therapy; 2) the spleen/liver, if considered enlarged due to lymphoma based on CT scan prior to therapy, would be normal and nodules should disappear; and 3) if bone marrow was involved before treatment, the infiltrate must clear on repeat bone marrow biopsy. Computed tomography (CT) scans of the neck, thorax, abdomen and pelvis were performed as part of the efficacy evaluation.
Time Frame: 200 weeks
Population: The Intent-to-treat (ITT) analysis set, comprised of all randomized participants, was analyzed.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Rituximab
Number analyzed (Participants) | 219 | 219
Participants | 36 | 44

3. Secondary Outcome: Number of Participants With Overall Response (OR)
Description: The overall response rate (ORR) was defined as the number of participants achieving a CR or partial response (PR). from start of randomization until disease progression, or the start of a new anti-cancer therapy. Disease response was assessed according to modified 2007 Revised Response Criteria for Malignant Lymphoma (RRCML). Computed tomography (CT) scans of the neck, thorax, abdomen and pelvis were performed as part of the efficacy evaluation. Bone marrow examination to confirm a suspected complete response (CR) was performed within 8 weeks following the onset of a CT scan confirmed CR.
Time Frame: 200 weeks
Population: The Intent-to-treat (ITT) analysis set, comprised of all randomized participants, was analyzed.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Rituximab
Number analyzed (Participants) | 219 | 219
Participants | 110 | 144

4. Secondary Outcome: Number of Deaths
Description: The number of deaths were assessed.
Time Frame: 200 weeks
Population: The Intent-to-treat (ITT) analysis set, comprised of all randomized participants, was analyzed.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Rituximab
Number analyzed (Participants) | 219 | 219
Participants | 28 | 30

5. Secondary Outcome: Number of Participants With Infection Related Adverse Events
Description: The number of participants with infection related adverse events was assessed.
Time Frame: 200 weeks
Population: The safety set, comprised of all participants who received one dose of study drug, was analyzed.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Rituximab
Number analyzed (Participants) | 217 | 218
Participants | 69 | 81

6. Secondary Outcome: Number of Participants With Infusion Related Adverse Events Due to Study Drug
Description: The number of participants with infusion related adverse events due to study drug was assessed.
Time Frame: 36 weeks + 60 days
Population: The safety set, comprised of all participants who received one dose of study drug, was analyzed.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Rituximab
Number analyzed (Participants) | 217 | 218
Participants | 178 | 112

7. Secondary Outcome: Number of Participants With Myelosuppression Adverse Events
Description: The number of participants with myelosuppression adverse events was assessed.
Time Frame: 200 weeks
Population: The safety set, comprised of all participants who received one dose of study drug, was analyzed.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Rituximab
Number analyzed (Participants) | 217 | 218
Participants | 24 | 41

8. Secondary Outcome: Duration of Response (DOR)
Time Frame: 200 weeks
Population: The analysis of this outcome was not performed due to the early termination of the study. Please see the brief summary of the protocol section for additional details.
Arm/Group | Ofatumumab | Rituximab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to Next Treatment
Time Frame: 200 weeks
Population: as for outcome 8
Arm/Group | Ofatumumab | Rituximab
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Pharmacokinetics
Time Frame: 70 weeks
Population: as for outcome 8
Arm/Group | Ofatumumab | Rituximab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ofatumumab | Rituximab
Serious Adverse Events (participants affected / at risk) | 38/217 | 37/218
Other Adverse Events (participants affected / at risk) | 177/217 | 150/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab (N=217) | Rituximab (N=218)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Otosclerosis (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lymph gland infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 5
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 3
Septic shock (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Poor peripheral circulation (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab (N=217) | Rituximab (N=218)
Neutropenia (Blood and lymphatic system disorders) | 6 | 16
Abdominal pain (Gastrointestinal disorders) | 12 | 7
Constipation (Gastrointestinal disorders) | 17 | 11
Diarrhoea (Gastrointestinal disorders) | 20 | 15
Nausea (Gastrointestinal disorders) | 19 | 16
Asthenia (General disorders) | 9 | 14
Chills (General disorders) | 8 | 13
Fatigue (General disorders) | 21 | 28
Pyrexia (General disorders) | 9 | 21
Nasopharyngitis (Infections and infestations) | 14 | 22
Upper respiratory tract infection (Infections and infestations) | 13 | 11
Infusion related reaction (Injury, poisoning and procedural complications) | 40 | 19
Alanine aminotransferase increased (Investigations) | 3 | 11
Neutrophil count decreased (Investigations) | 10 | 16
White blood cell count decreased (Investigations) | 12 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 11
Headache (Nervous system disorders) | 11 | 20
Insomnia (Psychiatric disorders) | 14 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 13
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 14
Rash (Skin and subcutaneous tissue disorders) | 42 | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 41 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.